CLINICAL TRIAL: NCT06214910
Title: ThiPhiSA: New Pathways to Prevention From Community TB Screening in South Africa
Acronym: ThiPhiSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Human Sciences Research Council (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Adrienne E Shapiro, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00018448; 1R21AI179276-01 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis; HIV I Infection
Keywords: Tuberculosis; TPT; 3HP; differentiated service delivery; multi-month dispensing
MeSH Terms: conditions — Tuberculosis | interventions — 9 alpha,11 alpha,15 alpha-trihydroxy-16-phenoxy-17,18,19,20-tetranorprosta-4,5,13-trienoic acid; rifapentine

STUDY DESIGN:
Intervention Model Description: Household-level randomization -- all individuals in a household will be randomized to the same study arm of medication delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational: Community-based TB preventive therapy (TPT) (Other): Participants in the community arm will receive a multi-month dispensing packet at enrollment with the complete 3 month supply of TPT (3HP: 3 months of weekly isoniazid and rifapentine).
  Interventions: Other: Community-delivered TB preventive therapy (TPT) - 3 months weekly isoniazid plus rifapentine (3HP)
- Standard-of-Care Tuberculosis Preventative Therapy (TPT) (Active Comparator): Participants in the standard of care arm will receive a referral letter to their local Department of Health (DoH) clinic to continue TPT. They will be instructed to present to the DoH clinic within 2 weeks to receive their continuation doses of TPT per current South African DoH standard of care (refills administered monthly).
  Interventions: Other: Clinic-link TPT

INTERVENTIONS:
Other: Community-delivered TB preventive therapy (TPT) - 3 months weekly isoniazid plus rifapentine (3HP) — Participants randomized to this arm will receive the entire supply of TB preventive therapy (TPT) at enrollment.
  Arms: Investigational: Community-based TB preventive therapy (TPT)
Other: Clinic-link TPT — Participants receive 2-week supply of TPT at initiation, then continue to receive remainder of TPT course at clinic (including refills).
  Arms: Standard-of-Care Tuberculosis Preventative Therapy (TPT)

SUMMARY:
This study will compare community-delivered, multi-month dispensing of tuberculosis preventive therapy (TPT) to standard-of-care clinic-based TPT delivery in a population of South African adults who are recommended to receive TB preventive therapy.

We hypothesize that persons receiving multi-month dispensing of TPT in the community will have a higher rate of TPT completion at 3 months than persons receiving TPT via standard of care with monthly clinic-based refills.

DETAILED DESCRIPTION:
The research objective is to understand and overcome key barriers to tuberculosis preventive therapy (TPT) delivery and completion in South Africa in the setting of 3HP scale-up. (3HP: short-course TPT consisting of 3 months weekly isoniazid[H] plus rifapentine [P]). The study will investigate these factors through a trial comparing community-delivered TPT, to clinic-based TPT and qualitative research investigating barriers to TPT completion and exploring task-shifted TPT delivery.

Aim 1: To determine the effect of community-based initiation and delivery of TPT on TPT completion.

Hypothesis: Community-delivered TPT will be associated with higher initiation and completion of TPT than standard of care clinic-based TPT.

Approach: Persons eligible for TPT will be identified through the Triage+ TB study and other community-based TB screening activities. Eligible persons will be randomized at the household level to 1) Immediate initiation of TPT & full 12 weeks delivery at once, or 2) Immediate initiation of TPT, 2-week supply, and referral to clinic for TPT completion. TPT adherence and completion will be measured by a combination of self-report, pill count, and serum drug level indicators.

Aim 2: To determine factors associated with TPT initiation and completion in people eligible for TPT identified in community settings.

Hypothesis: People with HIV (PWH) will have better rates of initiation and completion of TPT than people without HIV.

Approach: Participant interviews and surveys at baseline and end-of-study will assess willingness to take TPT, barriers and facilitators for individuals, experience taking TPT, and experience of interactions in clinic settings. Focus groups will be purposively selected based on end-of-study survey responses to elicit factors determining patient experience.

Aim 3: To determine feasibility and acceptability of differentiated service delivery (DSD) approaches, including task-shifting, for TPT delivery and scale-up.

Hypothesis: DSD TPT will be feasible and acceptable. Approach: Participatory qualitative research, and implementation science approaches including workflow mapping will be used to assess clinician-level barriers and inefficiencies in providing clinic-based TPT. In-depth interviews and focus groups will be conducted with pharmacy assistants, nurses, clinic operational managers, and district program managers to assess acceptability. Clinic flow will be mapped to determine effect of task-shifted pharmacy assistant TPT delivery on workflow and patient experience in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Living in the study catchment area
* Eligible for TPT according to South African National guidelines(5), i.e. are a) living with HIV or b) are a close contact of a person with TB disease (defined by a person that resides in the same house as a person with TB), c) and in either case
* Have screened negative for TB disease in the last 6 months, through TB TRIAGE+ Trial, other household contact tracing, or other community TB screening
* Negative TB screening at enrolment (if TB TRIAGE+ screening was more than 3 months ago)
* Willing and able to provide written or verbal consent
* Participants whom have not received TPT in the last 12 months; this was confirmed verbally with participants during the enrolment process.

Exclusion Criteria:

* Less than 18 years of age.
* Pregnant or planning on pregnancy within next three months
* Planning on moving or relocating from the area within the next three months
* Positive for active TB
* Currently on TB treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Completion of a course of TB preventive therapy (TPT) | 3 months, extended to 16 weeks as needed
  TPT completion defined as taking 11 doses of 3HP (3 months weekly isoniazid [H] plus rifapentine [P] ) within 16 weeks of 3HP initiation. The outcome will be measured as a composite outcome including: self-report of doses taken, periodic pill counts, one-time serum drug level of isoniazid.

SECONDARY OUTCOMES:
Overall adherence with TPT | 3 months, extended to 16 weeks as needed
  Proportion of doses completed
Predictors of TPT adherence | 3 months, extended to 16 weeks as needed
Participant satisfaction with the assigned TPT delivery method | 3 months, extended to 16 weeks as needed
  assessed by questionnaire
Adverse events | 3 months, extended to 16 weeks as needed
  Assessed by adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne E Shapiro, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Human Sciences Research Council, Sweetwaters, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Misra S, Madonsela T, Thomas KK, Grabow C, Lenn M, Morton JF, Reither K, Lynen L, van Heerden A, Essack Z, Bosman S, Shapiro AE. ThiPhiSA: new pathways to TB prevention from community screening - a household-randomised controlled trial in KwaZulu-Natal, South Africa. BMJ Open. 2025 Aug 12;15(8):e100927. doi: 10.1136/bmjopen-2025-100927. PMID 40803739